CLINICAL TRIAL: NCT00576498
Title: Detection Of Intestinal Metaplasia And High Grade Dysplasia In Barrett's Esophagus Using Novel Imaging Techniques - A Randomized Controlled Trial.
Brief Title: Novel Imaging Techniques in Barrett's Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency); Medical University of South Carolina (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, PRATEEK SHARMA, Professor of Medicine, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 00225(PS0036)
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Barrett Esophagus; Gastroesophageal Reflux
Keywords: GERD; NBI; AFI; IM; SSBE; LSBE; LGD; HGD
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1- Narrow Band Imaging (Experimental): NBI-AFI imaging - Narrow Band Imaging- Patients will be evaluated with a standard magnification endoscope (Olympus GIF Q240Z, 115x or GIF-H180 or equivalent) using a NBI light source.
  Autofluorescence Imaging (AFI)- Patients will be evaluated using a prototype autofluorescence endoscope (Olympus, Tokyo, Japan; excitation 395-475 nm, fluorescence detection 490-625 nm, red reflectance 600-620 nm and green reflectance 540-560 nm)
  Interventions: Other: NBI-AFI imaging
- 2-Standard Endoscopy (Other): Standard Endoscopy- Patients will undergo EGD with biopsies using a standard diagnostic video endoscope (Olympus, GIF 140 or 160) using the Seattle protocol - 4 quadrant biopsies using standard biopsy forceps every 2 cms; stored in separate jars
  Interventions: Other: Standard Endoscopy

INTERVENTIONS:
Other: NBI-AFI imaging — Narrow Band Imaging- Patients will be evaluated with a standard magnification endoscope (Olympus GIF Q240Z, 115x or GIF-H180 or equivalent) using a NBI light source.Target biopsies with standard biopsy forceps will be obtained from the different visualized patterns in separate jars.
  Autofluorescence Imaging- Patients will be evaluated using a prototype autofluorescence endoscope (Olympus, Tokyo, Japan; excitation 395-475 nm, fluorescence detection 490-625 nm, red reflectance 600-620 nm and green reflectance 540-560 nm).In this system, normal squamous and non-dysplastic BE appears green while the dysplastic areas appear magenta/purplish. Targeted biopsies will be obtained from the areas with abnormal fluorescence.
  Other Names: NBI; AFI
  Arms: 1- Narrow Band Imaging
Other: Standard Endoscopy — Standard Endoscopy- Patients will undergo EGD with biopsies using a standard diagnostic video endoscope (Olympus, GIF 140 or 160) using the Seattle protocol - 4 quadrant biopsies using standard biopsy forceps every 2 cms; stored in separate jars.
  Other Names: EGD
  Arms: 2-Standard Endoscopy

SUMMARY:
Primary Aim: In patients with endoscopically suspected BE, compared to standard endoscopy, novel techniques (NBI and AFI) with target biopsies will

* Detect more patients with intestinal metaplasia
* Detect more areas of high grade dysplasia
* Require fewer biopsies and a shorter time for procedure completion

Secondary Aim:

* Compare the yield of high-grade dysplasia(HGD)using NBI/AFI versus standard endoscopy with biopsy.
* Compare the number of biopsies and procedure times for NBI/AFI versus standard endoscopy with biopsy.
* Compare the inter-observer variability in classifying different mucosal and vascular patterns observed by NBI/AFI using kappa statistics.

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is the pre-malignant lesion for adenocarcinoma of the esophagus and esophagogastric junction. It is a condition in which the squamous mucosa of the distal esophagus is replaced by columnar mucosa, specifically intestinal metaplasia. The incidence of esophageal adenocarcinoma has been rapidly rising and has increased 3-6 fold over the past two decades. This has driven efforts to identify patients with the pre-malignant lesion i.e. BE. Intestinal metaplasia within the columnar lined esophagus is the epithelial type that predisposes patients to the development of adenocarcinoma; the other two epithelial types being cardiac and fundic.

Since intestinal metaplasia is now included in the definition and is the epithelial type associated with cancer, obtaining biopsies from the columnar lined distal esophagus is mandatory. The sensitivity and the positive predictive value of standard EGD for diagnosing BE has been reported as 82% and 34% respectively. This is secondary to the patchy and mosaic presence of intestinal metaplasia in the columnar distal esophagus. Endoscopic screening is advocated in patients with chronic GERD symptoms for detection of BE with random biopsies being obtained if a columnar appearing distal esophagus is visualized. Once intestinal metaplasia is detected with these random biopsies and the diagnosis of BE is confirmed, patients are subsequently enrolled in a surveillance program. Similarly, the presence of dysplasia or early adenocarcinoma within a segment of BE is patchy and focal and standard endoscopy and random biopsies may fail to detect these lesions. New endoscopic imaging techniques to improve the accuracy of endoscopic diagnosis have recently been developed, and most are currently under evaluation.

METHODS Study Overview:Patient presenting to GI lab for BE screening and surveillance Informed consent signed and patient randomized, if endoscopic BE is suspected to NBI target biopsies or standard endoscopy with biopsies as the first procedure If randomized to NBI first: patterns noted, target biopsies obtained from specific patterns Same patient returns in 3-6 weeks for 2nd procedure Standard endoscopy: 4 quadrant every 2 cms. random biopsies (i.e. standard BE surveillance) Findings of NBI and random biopsies compared after all patients complete protocol and results analyzed A process similar to the one outlined above will be used in comparing autofluorescence imaging to conventional endoscopy in patients with Barrett's mucosa.

Study Design:This study is part of a multicenter randomized controlled trial being conducted at two sites, the other one being Medical University of South Carolina. Patients will be randomized (opaque sealed envelopes generated by statistician) to undergo NBI/AFI or standard endoscopy with biopsies on day 1. The same patient will return for the alternative procedure with biopsies within 3-6 weeks of the 1st procedure and will be maintained on acid suppressive therapy during this time interval. Each patient will thus act as his/her own control. At the time of performing the 2nd procedure (either NBI/AFI target biopsies or standard endoscopy), the endoscopist will be blinded and will not be aware of the biopsy results from the 1st procedure. Every attempt will also be made to keep the endoscopists blinded to the past history of the patient i.e. non dysplastic BE, LGD, HGD etc.

Risk and benefit to the study participant:Data on newer imaging method like NBI and AFI are mostly in the form of case series. This has not led to a change in the standard of care. The early data is very encouraging but not conclusive due to lack of randomized, controlled trials. Hence, we chose a study design of randomized controlled trial of the newer modalities versus the existing conventional endoscopy. This design necessitates the performance of a repeat endoscopy. Upper endoscopy is very safe, routinely done procedure with a low risk of complications. A repeat procedure may, indeed, increase the potential for risks associated with the procedure but the magnitude is small. The added advantage of second endoscopy would be increased detection of dysplasia and adenocarcinoma resulting in potential benefit to the patients. The main reason for the performance of the current study is the limitation of conventional endoscopy with the implication that dysplasia and adenocarcinoma will be missed on the initial endoscopy. In clinical practice, this usually warrants a follow up endoscopy that is performed at 1-3 yr intervals due to time and cost constraints. For the study population of this trial, the second endoscopy has the potential for increased detection of dysplasia/early adenocarcinoma in the Barrett's segment that could lead to initiation of curative therapy.

Study Population:Patients undergoing BE screening and surveillance will be enrolled after written, informed consent. BE definition- columnar mucosa in the distal esophagus of any length with intestinal metaplasia on biopsy. The BE length will be measured from the gastroesophageal junction to the proximally displaced squamo-columnar junction. The patient demographics (age, gender and ethnicity) and the BE length will be recorded. Total time required for each procedure will be recorded - from endoscope insertion to removal.

Narrow Band Imaging: Patients will be evaluated with a standard magnification endoscope (Olympus GIF Q240Z, 115x or GIF-H180 or equivalent) using a NBI light source (already available at both centers). The outer diameter of the endoscope is 10.8 mm similar to standard diagnostic endoscopes. No special processing or cleaning of the endoscope is required - similar to the standard Olympus GIF-100. A cap may or may not be fitted on the distal tip of the endoscope allowing the mucosa in contact with the cap to be magnified without the motility of the esophagus affecting visualization. The different patterns will be grouped into ridge/villous, circular and irregular/distorted. Target biopsies with standard biopsy forceps will be obtained from the different visualized patterns in separate jars.

Autofluorescence Imaging: Patients will be evaluated using a prototype autofluorescence endoscope (Olympus, Tokyo, Japan; excitation 395-475 nm, fluorescence detection 490-625 nm, red reflectance 600-620 nm and green reflectance 540-560 nm). The AFI scope has two different CCD (charge coupled device to detect the light waves emitted/reflected from the biological tissue - similar to the chip used in a digital camera), one for conventional and another for AFI endoscopy. There is also a rotary filter that allows blue, red or green light to be generated selectively. The video processor constructs video images (AFI images or normal optical images) based on the signals provided by CCD at the distal end of the endoscope. In this system, normal squamous and non-dysplastic BE appears green while the dysplastic areas appear magenta/purplish. Targeted biopsies will be obtained from the areas with abnormal fluorescence. Both the NBI and AFI equipment will be supplied by Olympus America Inc.

Standard Endoscopy: Patients will undergo EGD with biopsies using a standard diagnostic video endoscope (Olympus, GIF 140 or 160) using the Seattle protocol - 4 quadrant biopsies using standard biopsy forceps every 2 cms; stored in separate jars.

Histology: All biopsy specimens will be stained with H&E and alcian blue at pH 2.5 & will then be reviewed by two pathologists (SM) and (DL), one at each site, who will be blinded to the NBI/AF results and patterns. Any disagreement in the histological diagnosis will be resolved by a consensus diagnosis. Dysplasia will be classified as no dysplasia, LGD, HGD and adenocarcinoma.

Data Collection:Patient demographics, order of randomization, endoscopy findings (BE length, NBI patterns, AFI patterns), procedure time, number of biopsies and histology reports will be collected and recorded by the study coordinator. All this information will be transferred into an ACCESS database

Statistical Power & Data Analysis:For the primary outcome, to determine if NBI/AFI target biopsies can diagnose BE (intestinal metaplasia) in 90% of the patients assuming that standard endoscopy with biopsy can diagnose Barrett's in 70%, we would need 122 patients in order to detect a significant difference between the two with 80% power and a type I error rate of 5% using McNemar's test for paired dichotomous responses.

For the secondary outcome of detection of HGD will be based on number of biopsies harboring HGD. If we assume that NBI/AFI can detect areas of HGD (within the BE segment) in 90% of the biopsies from irregular/distorted patterns compared to 60% by standard endoscopy, we would need to study 59 areas/biopsies of HGD in order to detect a significant difference between the two with 80% power and a type 1 error rate of 5% using McNemar's test for paired dichotomous responses. If we enroll at least 10-12 patients with HGD with an average BE length of 5 cms, we will be able to evaluate > 60 areas of HGD with each procedure. Each site will have to enroll approximately 30-35 BE patients (including 5-6 with HGD) each year.

McNemar's test will be used to compare paired categorical data while continuous paired data will be compared using non-parametric methods such as the Wilcoxon Sign Rank Test. A p value of <0.05 will be considered significant.

For the initial 30 consecutive patients enrolled in the study, inter-observer variability will be studied on the mucosal and vascular patterns and autofluorescence patterns.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected Barrett's esophagus on endoscopy
* Age > 18 years
* Ability to provide written informed consent

Exclusion Criteria:

* Presence of erosive esophagitis
* Visible nodules, lesions within Barrett's esophagus segment
* Endoscopist aware of biopsy results
* Inability to obtain biopsies due to anticoagulation or varices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with biopsy confirmed intestinal metaplasia | 08/2006 to 10/2008

SECONDARY OUTCOMES:
Detection of high grade dysplasia | 08/2006 to 10/2008
Procedure time | 08/2006 to 10/2008
Number of biopsies | 08/2006 to 10/2008
Inter observer variability in reading of mucosal and vascular patterns | 08/2006 to 10/2008

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Veterans Affairs Medical Center, Kansas City, MO; University of Kansas School of Medicine
Locations (3):
- United States (2):
  - Veterans Affairs Medical Center, Kansas City, Missouri
  - Medical University of South Carolina, Charleston, South Carolina
- Academisch Medisch Centrum-Universiteit van Amsterdam (AMC-UvA), Amsterdam, Netherlands

REFERENCES:
- [Background] Weinstein WM, Ippoliti AF. The diagnosis of Barrett's esophagus: goblets, goblets, goblets. Gastrointest Endosc. 1996 Jul;44(1):91-5. doi: 10.1016/s0016-5107(96)70239-0. No abstract available. PMID 8836727
- [Background] Devesa SS, Blot WJ, Fraumeni JF Jr. Changing patterns in the incidence of esophageal and gastric carcinoma in the United States. Cancer. 1998 Nov 15;83(10):2049-53. PMID 9827707
- [Background] Brown LM, Devesa SS. Epidemiologic trends in esophageal and gastric cancer in the United States. Surg Oncol Clin N Am. 2002 Apr;11(2):235-56. doi: 10.1016/s1055-3207(02)00002-9. PMID 12424848
- [Background] Gerson LB, Shetler K, Triadafilopoulos G. Prevalence of Barrett's esophagus in asymptomatic individuals. Gastroenterology. 2002 Aug;123(2):461-7. doi: 10.1053/gast.2002.34748. PMID 12145799
- [Background] Rex DK, Cummings OW, Shaw M, Cumings MD, Wong RK, Vasudeva RS, Dunne D, Rahmani EY, Helper DJ. Screening for Barrett's esophagus in colonoscopy patients with and without heartburn. Gastroenterology. 2003 Dec;125(6):1670-7. doi: 10.1053/j.gastro.2003.09.030. PMID 14724819
- [Background] Hamilton SR, Smith RR, Cameron JL. Prevalence and characteristics of Barrett esophagus in patients with adenocarcinoma of the esophagus or esophagogastric junction. Hum Pathol. 1988 Aug;19(8):942-8. doi: 10.1016/s0046-8177(88)80010-8. PMID 3402983
- [Background] Sampliner RE. Practice guidelines on the diagnosis, surveillance, and therapy of Barrett's esophagus. The Practice Parameters Committee of the American College of Gastroenterology. Am J Gastroenterol. 1998 Jul;93(7):1028-32. doi: 10.1111/j.1572-0241.1998.00362.x. No abstract available. PMID 9672324
- [Background] Sharma P, McQuaid K, Dent J, Fennerty MB, Sampliner R, Spechler S, Cameron A, Corley D, Falk G, Goldblum J, Hunter J, Jankowski J, Lundell L, Reid B, Shaheen NJ, Sonnenberg A, Wang K, Weinstein W; AGA Chicago Workshop. A critical review of the diagnosis and management of Barrett's esophagus: the AGA Chicago Workshop. Gastroenterology. 2004 Jul;127(1):310-30. doi: 10.1053/j.gastro.2004.04.010. PMID 15236196
- [Background] Eloubeidi MA, Provenzale D. Does this patient have Barrett's esophagus? The utility of predicting Barrett's esophagus at the index endoscopy. Am J Gastroenterol. 1999 Apr;94(4):937-43. doi: 10.1111/j.1572-0241.1999.990_m.x. PMID 10201460
- [Background] Inadomi JM, Sampliner R, Lagergren J, Lieberman D, Fendrick AM, Vakil N. Screening and surveillance for Barrett esophagus in high-risk groups: a cost-utility analysis. Ann Intern Med. 2003 Feb 4;138(3):176-86. doi: 10.7326/0003-4819-138-3-200302040-00009. PMID 12558356
- [Background] Cameron AJ, Carpenter HA. Barrett's esophagus, high-grade dysplasia, and early adenocarcinoma: a pathological study. Am J Gastroenterol. 1997 Apr;92(4):586-91. PMID 9128304
- [Derived] Sharma P, Hawes RH, Bansal A, Gupta N, Curvers W, Rastogi A, Singh M, Hall M, Mathur SC, Wani SB, Hoffman B, Gaddam S, Fockens P, Bergman JJ. Standard endoscopy with random biopsies versus narrow band imaging targeted biopsies in Barrett's oesophagus: a prospective, international, randomised controlled trial. Gut. 2013 Jan;62(1):15-21. doi: 10.1136/gutjnl-2011-300962. Epub 2012 Feb 7. PMID 22315471